CLINICAL TRIAL: NCT02066025
Title: Blood Test for Breast Cancer Associated Auto Antibodies - Improvement of Octava Blood Test
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Eventus Diagnostics Ltd (Industry)
Responsible Party: Sponsor
Other Study IDs: OctavaBreast_1
Record Dates: First submitted 2014-02-09; First posted 2014-02-19 (Estimated); Last update posted 2014-02-19 (Estimated); Status verified 2014-02

CONDITIONS: Breast Cancer
Keywords: breast cancer; cancer associated auto antibodies; breast cancer blood test
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Human plasma samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- group_0: Women with negative mammography (BIRADS 1-2), as negative controls.
- group_1: Women with positive biopsy for (ID, IL, DCIS) as patients.
- group_2: Women with positive mammography (BIRADS 3-4-5-6), and a negative biopsy diagnosis for breast cancer (ID, IL, DCIS) will be enrolled as benign (ADH, ALH, LCIS, fibroadenoma, fibrocystic changes (including sclerosing adenosis), Benign papillaoma, normal breast) as benigns.

SUMMARY:
Octava has two versions, each with a different intend of use.

OctavaPink is a qualitative in vitro diagnostic test service, performed by authorized clinical laboratories. The product is used for two following indications:

* Intend of Use #1: OctavaPink is indicated for women above 18 years old, who performed mammography and were determined negative for breast cancer. Being moderately sensitive (>55% sensitivity) the test is able to detect 55% of mammography false negatives. In addition, being highly specific (>95% specificity) it supplies additional evidence for true mammography negative result which will reduce examinees anxiety of being misdiagnosed as a result of high false negative mammography rate (10-30%)
* Intend of Use #2: OctavaPink is indicated for women above 18 years old, who performed biopsy after positive mammography and the biopsy result was negative. Being moderately sensitive (>55% sensitivity) the test is able to detect 55% of biopsy false negatives. In addition being highly specific (>95% specificity) it supplies an additional evidence for true biopsy negative result which reduces examinees anxiety of being misdiagnosed.

OctavBlue is a qualitative in vitro diagnostic test service, performed by EventusDx authorized laboratories. Intend of use of OctavBlue is the following:

• OctavBlue is indicated for women above 18 years old, who performed mammography and received doubtful results. Being highly sensitive (>95% sensitivity) the test can help to reveal 95% of positive cases; and being moderately specific (>55% specificity) - about half of negative cases. The test is not intended to be used as a standalone diagnostic technique but to supply additional information to a physician and help deciding about the further course of diagnosis.

DETAILED DESCRIPTION:
The primary objectives - To improve the specifications of the OctavaPink test and the OctavaBlue test. The current specifications being

1. For the OctavaPink - 95% specificity and 50% sensitivity.
2. For the OctavaBlue - 50% specificity and 95% sensitivity.

The study will be considered as successful in any of the below options -

1. If the new antigens incorporated in the OctavaPink chip will maintain specificity of at least 95% and increase the sensitivity to at least 85%.
2. If the new antigens incorporated in the OctavaBlue chip will maintain sensitivity of at least 95% and increase the specificity to at least 85%.

ELIGIBILITY:
Inclusion Criteria:

* Female subjects 18 years or over.
* Subjects following a mammography test.
* Subject with pathological evaluation after mammography with BIRADS 3-4-5-6.

Exclusion Criteria:

* Female Subjects less than 18 years of age
* Previous or concurrent malignancies
* Autoimmune disorders diagnosed subjects
* Hematological malignancies
* Subjects under active chemotherapy treatment or chemotherapy in the past 6 months
* Steroid treatment in the past 3 months
* Subject undergoing immunosuppressive treatments
* Subject with verified breast cancer other than invasive ductal or invasive lobular as verified by biopsy/cytology

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The target population will be any women with a mammography result (positive or negative).
  Women with negative mammography will be tested with the OctavaPink version to provide additional information to the doctors following a negative mammography.
  Women with a positive mammography will be tested with OctavaBlue version to provide additional information to a physician.
Sampling Method: Probability Sample
Enrollment: 1425 (Estimated)
Dates: Start 2014-03; Primary Completion 2016-03 (Estimated); Study Completion 2018-03 (Estimated)

PRIMARY OUTCOMES:
Number of participants in each of the clinicaly defined groups (0,1 and 2). | 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Galit Yahalom, Ph.D, Study Director — Eventus Dx
Locations (1):
- "Carmel" Medical Center, Haifa, Israel

REFERENCES:
- [Result] Yahalom G, Weiss D, Novikov I, Bevers TB, Radvanyi LG, Liu M, Piura B, Iacobelli S, Sandri MT, Cassano E, Allweis TM, Bitterman A, Engelman P, Vence LM, Rosenberg MM. An Antibody-based Blood Test Utilizing a Panel of Biomarkers as a New Method for Improved Breast Cancer Diagnosis. Biomark Cancer. 2013 Nov 19;5:71-80. doi: 10.4137/BIC.S13236. eCollection 2013. PMID 24324350